CLINICAL TRIAL: NCT06227299
Title: INTEGRAL Study: A Longitudinal Study of Surgeries and Lasers in Glaucoma: Long-term Results and Success Predictors Analysed From a Large-scale Retrospective and Prospective Glaucoma Register
Brief Title: INTEGRAL Study: A Longitudinal Study of Surgeries and Lasers in Glaucoma
Status: Enrolling by invitation | Type: Observational
Sponsor: Swiss Glaucoma Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: INTEGRAL
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Glaucoma patients: Patients with glaucoma

SUMMARY:
The aim of this study is to create a large-scale register of all glaucoma patients diagnosed, followed and treated in a large tertiary centre specialising in glaucoma, in order to analyse whether specific factors influence the progression of the disease or guide our choice of treatment. This should lead to a better understanding of the disease and the factors to be taken into account when choosing the best treatment option for each patient, leading to safer, more effective and patient-centred care.

DETAILED DESCRIPTION:
Glaucoma encompasses a group of chronic diseases characterized by progressive retinal nerve fibre loss and a concomitant pattern of visual field damage, eventually leading to blindness. To date, it is still considered the first cause of irreversible blindness worldwide. In recent years, treatment options for glaucoma have soared, and ophthalmologists can resort to a wide selection of drops, laser procedures and surgical techniques to reduce intraocular pressure, and slow the progression of the disease. The choice of the technique, however, often depends on personal preferences and it is still unclear if a specific technique is more efficient or safe, or if any patient-depending factors should guide the choice of treatment. The aim of this study is to create a large-scale register of all glaucomatous patients diagnosed, followed-up and treated in a large glaucoma-specialised tertiary centre, to analyse if any specific factor influence the progression of the disease or guide our treatment choice. This should lead to a better understanding of the disease itself and of the factors that should be considered when choosing the best treatment option for each patient, leading to safer, more efficient and more patient-centered care. This registry is thus of great importance for both patients and clinicians in the diagnosis and treatment of glaucoma.

The study is an observational analysis of patients' medical data recorded in a large-scale register, both retrospective and prospective.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of glaucoma (open-angle, closed-angle, primary or secondary) or ocular hypertension (IOP > 24 mmHg, medicated or not)
* Patients who received treatment (medical, laser or surgical) at the Glaucoma Centre, Montchoisi Clinic and Swiss Visio Montchoisi
* Age: 18 years old or older
* Able and willing to provide informed written or verbal consent

Exclusion Criteria:

* Patients who are unable to understand the implications of their inclusion in the study or who are unable or unwilling to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The register includes all patients diagnosed with glaucoma (primary, secondary, open and closed-angle) who received treatment at the Glaucoma Centre, at Montchoisi Clinic and Swiss Visio Montchoisi, Lausanne since 2014. There is no limit to the number of patients included in the register.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-05-29 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
IOP changes | 2 months, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  intraocular pressure (IOP) values compared to baseline
Number of molecules | 2 months, 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  • number of IOP-lowering medications required to maintain the IOP within therapeutic targets compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kaweh Mansouri, MD, Principal Investigator — Swiss Glaucoma Research Foundation
Locations (1):
- Swiss Visio Montchoisi, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No
IPD will be shared upon request from other researchers